CLINICAL TRIAL: NCT04816396
Title: The Effects of the Instrumental Reminiscence Therapy Based on Roy's Adaptation Model on Adaptation, Life Satisfaction and Happiness in Older Adults: A Randomized-controlled Trial
Brief Title: The Effects of the Instrumental Reminiscence Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Özlem Aydoğdu, PhD Candidate, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: eastern mediterranean
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Elderly; Reminiscence Therapy
Keywords: elderly; reminiscence Theraphy; Roy Adaptation Model; Nursing

STUDY DESIGN:
Intervention Model Description: Data Collection Process of Phase 1 of the Study In the 1st stage of this research; It is aimed to reveal the experiences of elderly people who have moved from their homes to nursing homes for the first time, regarding their adaptation to nursing homes. The results to be obtained will form the basis for the second phase of the research.
  The data will be collected by face-to-face interview method in depth in accordance with the qualitative research design. The interviews will be recorded with a tape recorder after the written and verbal consent of the participants. The talks will be held in a quiet and comfortable environment. The research will cease when the same information is started to be repeated by family members. Audio recordings will be destroyed after the data are analyzed.
  The research was planned to be conducted in an experimental type with pre-test and post-test control group.
Masking Description: In the first week of the study, Life Satisfaction Scale, Adaptation Scale, Diagnostic Form and Happiness Scale will be filled in. After 8 weeks of recall therapy, the scales will be re-evaluated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): For 8 weeks, Reminiscence Therapy based on Roy Adaptation Model will be applied
  Interventions: Behavioral: reminiscence Therapy
- No İntervention (No Intervention): No intervention will be applied to this group.

INTERVENTIONS:
Behavioral: reminiscence Therapy — Application Stages of Reminiscence Therapy Based on Roy Adaptation Model Week 1 (Session 1):Introduction-Meeting-Infancyand Family Life Week 2 (Session 2):Childhood and School Years Week 3 (Session 3):Unforgettable Historical Periods,Old movies, Old Songs Week 4 (Session 4):Loved, meals,Desserts and Recipes,Nutrition Style Week 5 (Session 5):Work and Marriage Week 6 (Session 6):Home and Garden Works,Animals, Plants Week 7 (Session 7): Travels, Vacation Memories Week 8 (Session 8): Celebration Memories, Evaluation Posttest Closing.
  Arms: experimental

SUMMARY:
This study was planned to determine the effect of Remembrance Therapy Based on Roy's Adaptation Model on the level of life satisfaction, harmony and happiness of the elderly. The research will be conducted with elderly individuals staying in Kalkanlı Yaşam Evi and Bülent Ecevit Rehabilitation Center. The research consists of 2 stages. In the first phase, the adaptation experiences of the elderly individuals who have been hospitalized in both institutions in the last year in a qualitative design, the results to be determined will form the basis of the second phase of the study. The second stage of the research is planned to be conducted in an experimental type with pre-test and post-test control group. The intervention group will be the elderly living in Kalkanlı Yaşam house, and the control group will be the elderly staying in Bülent Ecevit R. The elderly who are in the intervention group will be given Remembering Therapy once a week for a total of 8 weeks. In the study, the Standardized Mini Mental Test prepared by the researcher, the "Descriptive Information Form for the Elderly Person", which includes questions about sociodemographic, social and medical characteristics and aims to identify elderly individuals, and in addition to these, the "Happiness Scale" to determine the happiness level of the elderly individuals. ', "Life Satisfaction Scale" will be used to evaluate life satisfaction and "Elderly Adaptation Difficulty Scale" will be used to evaluate their adaptation. Data will be collected by the researcher through face-to-face interviews with the elderly

DETAILED DESCRIPTION:
The population of the elderly is increasing all over the world and in our country Globally, the number of people aged 65 and over is reported to be 727 million in 2020. In the next thirty years, it is predicted that the number of elderly people in the world will be over 1.5 billion and the rate of the population aged 65 and over, which was 9.3% in 2020, will increase to 16.0% in 2050. With the aging society, there are more elderly people in the service area of nurses. For this reason, there is a need to plan nursing interventions to improve and maintain elderly health and quality of life. With the increase of the elderly population in the world and in our country, the problems experienced by the elderly gain importance, and the necessity of interventions to meet their social and emotional needs comes to the fore.

The Roy Adaptation Model (RAM), developed by Sister Callista Roy, from an expanded, integrated and holistic nursing perspective (RAM), enables the development of theory-based nursing interventions in the process of adapting to old age and coping with the problems encountered. According to RAM, nursing balances knowledge of biology and behavioral sciences with "the understanding of individuals as both a physiological being in a physical world and as a creature that thinks and feels with human experience in a cosmic world. According to Roy, the general purpose of nursing is to improve the health of individuals and groups by enabling them to adapt to each of the four areas of adaptation, including physiological, self-concept, role function and interdependence. According to Roy, nurses contribute to improving the health of individuals and groups, as well as increasing the quality of life and dying in dignity. The elderly population is one of the groups that need adaptation. it is a process that requires adaptation to critical conditions of life such as separations, losses and approaching the end of life. Compliance is considered important in this age group. When elderly individuals cannot adapt to the aging process, they face some psychological problems such as loneliness, unhappiness, despair, loneliness, depression, and fear of death. This situation negatively affects the quality of life and life satisfaction of elderly individuals. In old age, with the increasing longing for the old, adaptation due to aging decreases, and the situation becomes difficult to cope with the addition of forgetfulness.

Recall therapy, which is used to cope with forgetfulness in elderly individuals, is one of the non-pharmacological approaches preferred in recent years for successful agin. It can significantly affect their ability to adapt. Recall therapy, in the Classification of Nursing Interventions (NIC), includes "remembering past events, feelings, and thoughts;" pleasure, quality of life or using it to facilitate adaptation to existing conditions ". In this context, reminiscence therapy takes an important place in nursing care as a therapeutic nursing intervention in order to increase the quality of life of the elderly and facilitate their adaptation processes.

Life satisfaction, which is an important element of quality aging, consists of basic indicators such as length of life, biological and mental health, cognitive competence, social competence, productivity, personal control and enjoyment of life. It has been stated that health-enhancing behaviors play an important role in increasing the life satisfaction of elderly individuals. In this context, group activities with the elderly; It enables the individual to keep his / her relationships with his / her social environment alive, to make efforts to improve memory and physical functions by bringing his creativity to the forefront, to look positively to life and to enjoy life Older participants in Aberg's qualitative study stated that their activity and independence are very important for their life satisfaction and that good past memories are remembered in this process. These health-enhancing reminiscence-based activities have an important place in reducing the years lost due to premature deaths, adding the remaining years to a healthy life and increasing life adaptation. is a process. Another concept related to the concept of satisfaction with life and positive on the quality of life is the concept of "happiness." Changes in old age and changes in lifestyle affect the happiness levels of the elderly. Happiness is an important indicator of well-being and healthy aging The concept of happiness is addressed with the concept of subjective well-being, and subjective well-being is defined as an individual's personal assessment of his life and reporting his own judgment. In the study of Akyıl et al., It was stated that those living at home and those who felt 'well' physically and psychologically had higher levels of subjective happiness.

In a study conducted, it was stated that there was a positive correlation between the autonomy level and happiness levels of elderly individuals, their happiness decreased and depression increased as their autonomy decreased. In another study conducted with the elderly living in institutions, 49.7% of the participants felt themselves unhapp .

Remember-based activities play a positive role in improving the quality of life of the elderly. In the literature, it is seen that studies examining the effects of reminiscence therapy on elderly health are often on quality of life, anxiety, and depression In the study of Tribe (2018), it is stated that reminiscence therapy has a positive effect on the sleep quality of the elderly living in institutions. and it is aimed to determine the effect on their happiness. It is thought that the results to be obtained will contribute to the planning of education and care activities aimed at improving the health of the elderly for health professionals working in institutions where elderly care services are provided. In this study, it is important to know the factors that affect the adaptation of the elderly first in planning the remembering therapy to be applied to the elderly. Therefore, the research will be conducted in two stages. The first phase will be carried out in accordance with the qualitative research design in order to reveal the life experiences related to the adaptation of the elderly who have transferred to the nursing home for the first time in the last year. In the second stage, it is aimed to determine the effect of reminiscence therapy based on the Roy Adaptation Model on the level of adaptation, life satisfaction and happiness of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Must be 65 years or older
* Should not have alzheimer schizophrenia or similar mental health problems
* Must be staying in nursing home

Exclusion Criteria:

* Willing to leave work voluntarily
* Not attending at least 3 interviews

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Adaptation Difficulty Rating Scale for the Elderly (YUGDÖ) | 6 mounth
  It is a 4-point Likert-type scale consisting of 24 items, which was developed by Şişman and whose validity and reliability were made to determine the adequacy of elderly individuals in adapting to old age. The scale items were determined as 0 points for "none" response, 1 point for "a little", 2 points for "quite" and 3 points for "a lot". In the scoring of the scale, the scores obtained from the items are calculated by adding up and dividing by the number of questions. The average score that can be obtained from the scale is the lowest 0, the highest 3. As the individual's score on the scale increases, the level of adaptation to old age decreases. Permission was obtained by e-mail for the use of the scale.
Life Satisfaction Index A / Life Satisfaction Scale Life Satisfaction Index A / Life Satisfaction Scale | 6 mounth
  It was developed by Neugarten et al. (1961) to measure the attitude to life and life satisfaction levels of elderly individuals. Its validity and reliability in Turkish society was also made by Karataş (1988). The scale consists of 20 questions consisting of yes / no options that measure individuals' view of different aspects of life, and how they perceive themselves and their environment, and is evaluated over 20 points. High scores indicate high life satisfaction. A scale score of 7 or below is considered to be a low life satisfaction level, a medium between 8-12, and a high level of satisfaction with life when it is 13 and above. Each option in the scale reflects 1 point, and some of the statements (3,5,7,10,14,17,18,20) should be answered no. Permission was obtained by e-mail for the use of the scale.
Oxford Happiness Scale Short Form | 6 Mounth
  It was developed by Hills and Argyle in 2002. Its Turkish translation and validity and reliability study was conducted by Doğan and Akıncı Çötok in 2011. The scale consists of 7 items and is in 5-point Likert type. Items 1 and 7 are coded in reverse. Permission was obtained by e-mail for the use of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Aydoğdu, 1, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean Universty, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis
Supporting Information: SAP, CSR
Time Frame: Unlimited use after September 2022
Access Criteria: No criteria, anyone can use

REFERENCES:
- [Result] Amieva H, Robert PH, Grandoulier AS, Meillon C, De Rotrou J, Andrieu S, Berr C, Desgranges B, Dubois B, Girtanner C, Joel ME, Lavallart B, Nourhashemi F, Pasquier F, Rainfray M, Touchon J, Chene G, Dartigues JF. Group and individual cognitive therapies in Alzheimer's disease: the ETNA3 randomized trial. Int Psychogeriatr. 2016 May;28(5):707-17. doi: 10.1017/S1041610215001830. Epub 2015 Nov 17. PMID 26572551
- [Result] Wu LF. Group integrative reminiscence therapy on self-esteem, life satisfaction and depressive symptoms in institutionalised older veterans. J Clin Nurs. 2011 Aug;20(15-16):2195-203. doi: 10.1111/j.1365-2702.2011.03699.x. Epub 2011 Jun 1. PMID 21631615
- [Result] Roy C, Whetsell MV, Frederickson K. The Roy adaptation model and research. Nurs Sci Q. 2009 Jul;22(3):209-11. doi: 10.1177/0894318409338692. No abstract available. PMID 19694080
- [Result] Rogers C, Keller C. Roy's adaptation model to promote physical activity among sedentary older adults. Geriatr Nurs. 2009 Mar-Apr;30(2 Suppl):21-6. doi: 10.1016/j.gerinurse.2009.02.002. No abstract available. PMID 19345860
- [Result] Wagner C, van der Wal G, Groenewegen PP, de Bakker DH. The effectiveness of quality systems in nursing homes: a review. Qual Health Care. 2001 Dec;10(4):211-7. doi: 10.1136/qhc.0100211... PMID 11743149